CLINICAL TRIAL: NCT06796881
Title: Instrument Assisted Soft Tissue Mobilization Versus Myofascial Release in Patients With Chronic Non¬Specific Low Back Pain
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Dalia Salah Ahmed elshatoury, principal investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Dalia-003373
Record Dates: First submitted 2025-01-22; First posted 2025-01-28 (Actual); Last update posted 2025-01-28 (Actual); Status verified 2025-01

CONDITIONS: Myofascial Release; Instrument Assisted Soft Tissue Mobilization; Chronic Low-back Pain
MeSH Terms: interventions — Myofascial Release Therapy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Instrument assisted soft tissue mobilization group (Experimental): treatment group A involved 22 patients who will receive instrumental-assisted soft tissue mobilization and exercises
  Interventions: Other: Instrument assisted soft tissue mobilization; Other: The conventional exercise program
- Myofascial Release group (Active Comparator): treatment group B involved 22 patients who will receive myofascial release and exercises
  Interventions: Other: Myofascial release; Other: The conventional exercise program
- Exercise only group (Active Comparator): control group (C) involved 22 patients who will receive exercises only.
  Interventions: Other: The conventional exercise program

INTERVENTIONS:
Other: Instrument assisted soft tissue mobilization — The group will undergo Instrument assisted soft tissue mobilization using M2Tblade, applying it for 40-120 seconds until hyperemia occurs. After treatment, ice packs will be applied for 5 minutes to reduce hyperemia. The therapist will ensure comfort through continuous communication and reporting any discomfort.
  Arms: Instrument assisted soft tissue mobilization group
Other: Myofascial release — The therapist will use a cross-hand release technique to release the lumbar spine, ensuring the patient is prone and suitable. They will lean into the patient to the tissue depth barrier, wait, and follow each release, avoiding force or slipping. The technique will be applied for 5 minutes on each side.
  Arms: Myofascial Release group
Other: The conventional exercise program — Patients will undergo a 12-session exercise program for 6 weeks, consisting of straight leg raising, bridging exercise, prone hip extension exercise, and abdominal curl exercise. The exercises will be done 3 sets, 10 repetitions each, with 1 minute rest between each set. The abdominal curl exercises involve supine or hook-lying positions with the lumbar spine neutral, with the patient performing a drawing in maneuver to stabilize the abdominal muscles. The progression involves lifting the shoulders, changing arm positions, and holding a weight or medicine ball. The patient's position is hook-lying, maintaining a neutral spinal position.

SUMMARY:
This study was done to compare the effect of instrumental-assisted soft tissue mobilization versus the effect of myofascial release on pain intensity, pressure pain threshold, back function, and back range of motion in patients with chronic nonspecific low back pain.

DETAILED DESCRIPTION:
Low back pain affects 20% of the workforce annually, leading to increased work absenteeism. Chronic non specific low back pain restricts functional and occupational activities, impacting society and the economy. Treatment is often unsatisfactory, and there is no consensus on the optimal approach. Further scientific research is needed to understand the effects of facial tissue manipulation on Chronic non specific low back pain patients. The literature has not addressed the distinctions between myofascial force transmission instrumental assisted soft tissue mobilization and myofascial release on Chronic non specific low back pain patients, which could help physical therapists find effective treatments. This study is the first to include pain, Pressure pain threshold, back function, and range of motion as outcome measures and compare instrumental assisted soft tissue mobilization and myofascial release in Chronic non specific low back pain patients.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with chronic non-specific low back pain for more than 3 months.
2. Age between 25-45 years.

Exclusion Criteria:

1. Patients who have serious spinal pathologies, such as fractures, tumors or inflammatory diseases (such as ankylosing spondylitis)
2. Patients who have nerve root compromise, disk herniation, spondylolisthesis with neurological involvement, or narrowing of spinal canal
3. Pregnant women
4. Cancer patients .
5. Lower limb injuries.
6. Body mass index (BMI) greater than 25.

Ages: 25 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 66 (Estimated)
Dates: Start 2025-01-23 (Actual); Primary Completion 2025-05-23 (Estimated); Study Completion 2025-06-24 (Estimated)

PRIMARY OUTCOMES:
Assessing the change of pain intensity using visual analogue scale | at baseline and after 6 weeks
  The visual analogue scale is a reliable tool for assessing chronic musculoskeletal pain, including chronic low back pain, with high correlations with verbal descriptive and numeric rating scales. It is a 10-cm line marked with no pain and severe pain, with higher scores indicating greater pain intensity.

SECONDARY OUTCOMES:
Assessing the change of pressure pain threshold using the pressure algometer | at baseline and after 6 weeks
  A 1-cm diameter disk with a calibrated dial gauge is used to measure soft tissue tenderness on myofascial trigger points. The force applied to the point gradually increases, and patients are instructed to stop the algometry when experiencing a painful sensation. The force in Pascal is then read from the display.
Assessing the change of flexion range of motion of the lumbar spine using the back range of motion device | at baseline and after 6 weeks
  The back range of motion II uses two Universal Inclinometers to measure range of motion to the spine, eliminating errors associated with stand-alone inclinometers. The investigator uses these inclinometers for flexion measurements, with the patient in an upright position. The therapist palpates and marks S1 and T12 on bare skin, centers the inclinometers, zeros them, and records the readings after the patient flexes forward.
Assessing the change of extension range of motion of the lumbar spine using the back range of motion device | at baseline and after 6 weeks
  The back range of motion II uses two Universal Inclinometers to measure range of motion to the spine, eliminating errors associated with stand-alone inclinometers. The investigator uses these inclinometers for extension measurements, with the patient in an upright position. The therapist will repeat flexion protocol for extension having the patient extends back for full extension and will record the value
Assessing the change of lateral flexion range of motion of the lumbar spine using the back range of motion device | at baseline and after 6 weeks
  The therapist will position the patient against a wall to prevent bending during lateral flexion measurements. The back range of motion unit will be adjusted until the inclinometer reads zero. For right lateral flexion, the patient will slide their hand down their leg while keeping their legs straight.
Assessing the change of rotation range of motion of the lumbar spine using the back range of motion device | at baseline and after 6 weeks
  The therapist will place the back range of motion unit, so the unit's feet are in line with T12. The therapist will hold the center of the unit firmly against the patient's back and zero the compass. The therapist will have the patient slowly turn the shoulders to either side, making sure they go to full range and record the reading
Assessing the change of back function using the 5) The Arabic version of Oswestry Disability Index | at baseline and after 6 weeks
  The Oswestry Disability Index is a self-reported questionnaire with 10 questions assessing daily living activities in patients with low back pain. The questions range from pain intensity to personal care and are scored on a 6-item Likert scale. The Arabic version of the oswestry disability index has good intra-observer reliability and good construct validity, with strong correlations with the visual analogue scale pain scale, Roland-Morris Low Back Pain Disability, and Quebec Back Pain Disability Scale.

CONTACTS AND LOCATIONS:
Locations (1):
- the Outpatient Clinic of the Police Authority Hospital, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No